CLINICAL TRIAL: NCT06754540
Title: Efficacy and Safety of Azacitidine Combined with Donor Lymphocyte Infusion for Prevention of Recurrence After Haploid Hematopoietic Stem Cell Transplantation in High-risk Acute Myeloid Leukemia
Brief Title: Azacitidine Combined with Donor Lymphocyte Infusion for Acute Myeloid Leukemia Post-transplant Relapse Prevention.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHSYXY-202405-AZA-DLI
Record Dates: First submitted 2024-12-29; First posted 2025-01-01 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia (AML); Relapse
Keywords: azacitidine; donor lymphocyte infusion; HSCT; haploid; high-risk; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AZA-DLI for acute myeloid leukemia post-transplant relapse preventiont (Experimental): One arm,Azacitidine is administered subcutaneously at 32 mg/m2/d for five consecutive days, starting no earlier than day +90 after HSCT, then repeated every 28 days for a total of twelve cycles. DLI is administered after an interval of 48 hours. Prophylactic DLI is given in escalating doses every four to six weeks for a total of three to four doses.The initial dose of DLI for haploid transplant patients is 1×10^5 CD3+/kg receptor weight lymphocytes gradually increased to 5×10^5, 1×10^6 and (2~5)×10^6 CD3+ Lymphocytes
  Interventions: Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: Azacitidine (AZA) — Azacitidine 32mg/m2

SUMMARY:
This study is single-center, single-arm, prospective, Phase II clinical trial with the primary objective of assessing the effectiveness of azacitidine combined with donor lymphocyte infusion (DLI) in the prevention of recurrence after high-risk haploid hematopoietic stem cells of AML.

At the screening/baseline period, informed consent is obtained and the inclusion/exclusion criteria are checked. Plan to enroll 51 patients, and collect demographic data, medical history data, vital signs, physical examination and laboratory tests (blood routine; urine routine; liver and kidney function;Immune indicators: T cell subsets, Treg, etc.), pregnancy tests for female patients and other necessary auxiliary inspections.The time to start treatment is from the +90 to +180 days after high-risk AML haploid hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
1.Basic solution: Azacitidine is administered subcutaneously at 32 mg/m2/d for five consecutive days, starting no earlier than day +90 after HSCT, then repeated every 28 days for a total of twelve cycles. DLI is administered after an interval of 48 hours. Prophylactic DLI is given in escalating doses every four to six weeks for a total of three to four doses.The initial dose of DLI for haploid transplant patients is 1×10^5 CD3+/kg receptor weight lymphocytes gradually increased to 5×10^5, 1×10^6 and (2~5)×10^6 CD3+ Lymphocytes.

1. Start time of medication: +90 ~ +120 days after transplantation.
2. Donor lymphocyte infusion was preceded by anti-anaphylaxis,such as promethazine and hormone therapy was prohibited.
3. In the course of AZA and DLI intervention, other targeted drugs such as venetoclax or chemotherapy drugs can be added on the basis of AZA if MRD or MRD increase (>1log) ,DLI continues as planned.

2.Stop treatment: Occurrence of any of the following conditions:

1. Life-threatening complications.
2. Acute GVHD above II degree; chronic GVHD above moderate manifestations or overlapping syndrome; No chronic GVHD is observed if acute GVHD remission is observed after discontinuation for 1 to 2 months, then preventive treatment is started again .
3. Hematologic recurrence, graft rejection or bone marrow donor chimerism <90%.

ELIGIBILITY:
Inclusion Criteria:

-

Patients enrolled must meet the following criteria:

1. ≥18 years old and ≤70 years old, male or female;
2. Patients with haploid peripheral blood stem cell transplantation of AML;
3. All patients received BU based myeloablative conditionings;
4. A diagnosis of high-risk AML is one of the following:

   ① Patients without morphologic CR before transplantation, including patients with initial refractory disease and recurrence.

   ② AML with poor prognosis (Standardized diagnosis and prognostic stratification of acute myeloid leukemia based on ELN edition which was 2022 Year) .
5. Blood routine: neutrophils ≥1×10^9/L, platelet ≥50.0×10^9/L;
6. There is no active grade II or higher acute GVHD or moderate or severe chronic GVHD;
7. The ECOG score is 0 to 2;
8. Donor lymphocytes are available;
9. The patient must be able to understand and be willing to participate in the study and sign an informed consent form.

Exclusion Criteria:

* Possible subjects who meet any of the following criteria will be excluded from the trial:

  1. Those who are allergic to known azacitidine or interferon
  2. Patients with active acute GVHD;
  3. Patients with moderate or more chronic GVHD;
  4. Non-haploid donor transplants;
  5. Patients who have not achieved complete remission after transplantation;
  6. AML recurrence after transplantation (bone marrow, peripheral blood primitive cells ≥5% or extramedullary recurrence), or graft rejection, bone marrow donor cell chimeric rate (STR) <90%;
  7. Patient blood routine: ANC<1.0×10^9/L or PLT<50×10^9/L;
  8. Combined with severe organ dysfunction:liver function (AST/ALT) >3 times normal upper limit; the direct bilirubin > 3 times normal upper limit; renal function (Cr) < 50mL/min or >1.5 times normal upper limit, regardless of hemodialysis treatment;
  9. Patient with severe active infection;
  10. Pregnant or lactating women;
  11. Have received other interventions or are receiving other research drugs before the study begins;
  12. At the discretion of the investigator, other dangerous complications may result.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Leukemia-free survival (LFS) time | From the date of transplantation, assessed up to 1 year after transplantation.
  Summary statistics for LFS time will be computed for all patients.

SECONDARY OUTCOMES:
overall survival (OS) | From the date of transplantation, assessed up to 1 year after transplantation.
  The method of Kaplan and Meier will be used to estimate the distribution of overall survival. Cox proportional hazards regression analysis will be used to model the association between overall survival and covariates of interest.
Cumulative incidence of relapse (CIR) | From the date of transplantation, assessed up to 1 year after transplantation.
  Use the method of Gooley et al to estimate the cumulative incidence of relapse.
Cumulative incidence of acute and chronic GVHD | From the date of transplantation, assessed up to 1 year after transplantation.
  Patients diagnosed with acute and chronic GVHD were recorded after DLI intervention.The definition of acute GVHD by national Institutes of Health (NIH) divides acute GVHD into classical acute GVHD and delayed acute GVHD
NRM | NRM
  The proportion of transplant-related deaths was recorded.
Incidence of toxicity of the regimen | From the date of transplantation, assessed up to 1 year after transplantation.
  Descriptive statistics will be used to summarize adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No